CLINICAL TRIAL: NCT03085524
Title: The Impact of Diabetes on REvascularization
Acronym: TIDE
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Carelon Research (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joshua Beckman, Professor, Vanderbilt University Medical Center
Other Study IDs: 161402
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Arterial Disease; Diabetes Mellitus
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Leukocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical Bypass: Subjects in the BEST-CLI trial assigned to surgical revascularization.
  Interventions: Diagnostic Test: Platelet function testing; Diagnostic Test: Vascular ultrasonography
- Endovascular: Subjects in the BEST-CLI trial assigned to endovascular revascularization.
  Interventions: Diagnostic Test: Platelet function testing; Diagnostic Test: Vascular ultrasonography

INTERVENTIONS:
Diagnostic Test: Platelet function testing — The investigators will test platelet reactivity at the beginning and midpoint of the first year after revascularization
Diagnostic Test: Vascular ultrasonography — The investigators will test bypass graft and stent patency at 30 days, 6 months, and 1 year.

SUMMARY:
The presence of foot symptoms at rest or tissue necrosis in patients with peripheral artery disease is a medical urgency and represents a state of critical limb ischemia (CLI) where the risk of amputation, in the absence of revascularization, is high. No trial conducted to date in peripheral revascularization has determined the effect of diabetes on mechanism of revascularization failure. Therefore, this trial represents a unique opportunity to investigate the mechanisms by which diabetes affects surgical and endovascular revascularization procedures with the long-term goal of improving outcomes in CLI.

DETAILED DESCRIPTION:
Peripheral artery disease is a condition defined by marked accumulation of atherosclerotic plaque below the distal aorta that reduces lower limb arterial perfusion. Blood flow reductions may be inadequate for exercising limbs and cause ischemic muscle pain, called intermitted claudication, or, in severe cases, the reduction may be inadequate for basal metabolism and cause pain at rest, ulceration, or gangrene. The presence of symptoms at rest or tissue necrosis is a medical urgency and represents a state of critical limb ischemia (CLI) where the risk of amputation, in the absence of revascularization, is high. The ageing of the population and the increasing prevalence of diabetes mellitus ensures this population will continue to grow in the foreseeable future. The impact of diabetes, however, is not limited to PAD incidence. Diabetic patients represent a particularly vulnerable subset of PAD patients and have a four-fold risk of CLI compared to non-diabetic patients. Indeed, in previous studies of CLI, more than half of patients have diabetes. As a result, the combination of diabetes and PAD accounts for more than half of non-traumatic amputations in the United States. Diabetic patients often present with foot ulcerations as their first manifestation of PAD and have challenging anatomy for revascularization. Failed vascular reconstructions, both endovascular or surgical, often result in additional tissue loss and transtibial amputations. Despite these challenges, the mechanisms of restenosis and the impact of diabetes have not been well explored for both types of revascularization in patients with CLI. The BEST-CLI trial is a multi-center, randomized, comparative effectiveness trial comparing open surgical bypass therapy to endovascular therapy in CLI patients with a composite clinical endpoint denoted as Major Adverse Limb Event free survival (MALE-free survival). However, the BEST-CLI trial does not study the mechanisms by which revascularization may fail. This proposal will extend the novel clinical work of the BEST-CLI trial by studying the mechanisms of bypass vein graft and stent failure. The investigators will adjudicate the mode of revascularization (vein graft or stent) in a central core laboratory, measure systemic markers of diabetic dysmetabolism including inflammation, insulin resistance, adverse adipokine expression, poor nutrition, and renal dysfunction, and begin to study the association of these factors with graft failure. Indeed, no trial conducted to date in either coronary or peripheral revascularization has determined the mechanism of revascularization failure, the impact of diabetes, nor the relationship between conduit patency and clinical outcomes. Therefore, this trial represents a unique opportunity to investigate the mechanisms by which diabetes affects surgical and endovascular revascularization procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 35 years or older
* Atherosclerotic, infrainguinal PAD
* CLI, defined as arterial insufficiency with gangrene, non-healing ischemic ulcer, or rest pain, consistent with Rutherford classes 4-6
* Candidate for either open or endovascular infrainguinal revascularization as judged by the treating investigators
* Adequate inflow into the index femoral artery
* Adequate popliteal, tibial, or pedal revascularization target
* Willing to comply with protocol, attend follow-up appointments, complete all study assessments, and provide informed consent
* Endovascular revascularization with a stent
* Surgical revascularization with a vein graft-

Exclusion Criteria:

* Femoropopliteal disease pattern consistent with TASC IIA
* Complete occlusion of the iliac artery
* Aortoiliac occlusive disease or severe common femoral artery disease
* Presence of a femoral, popliteal or tibial aneurysm of the index limb
* Life expectancy less than 2 years
* Deemed excessive risk for surgical bypass
* A vascular disease prognosis that includes an anticipated above ankle amputation on index limb within 4 weeks of index procedure
* Renal dysfunction defined as MDRD eGFR ≤ 30ml/min/173 m2 at the time of screening
* Currently on dialysis or history of a renal transplant
* A documented hypercoagulable state
* Nonatherosclerotic occlusive disease
* Any prior infrainguinal revascularization
* Current immuno-suppressive medication, chemotherapy or radiation therapy
* Absolute contraindication to iodinated contrast

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This ancillary study is an observational study design examining the effects of diabetes mellitus on restenosis following surgical or endovascular revascularization in CLI patients. Eligible patients will be screened according to the specified exclusion and inclusion criteria of the BEST-CLI trial.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Major Adverse Limb Event - free survival | 1 year
  The combination of amputation, surgical revascularization, thrombectomy, thrombosis, interposition graft, or death
Restenosis | 1 year
  Greater than 50% stenosis as determined by peak systolic velocity ratio of >2.4

CONTACTS AND LOCATIONS:
Locations (43):
- United States (38):
  - Long Beach VA Medical Center, Long Beach, California
  - Keck Medical Center of USC, Los Angeles, California
  - San Francisco VA Medical Center, San Francisco, California
  - University of California San Francisco Medical Center, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Loyola University Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Iowa Heart Center, West Des Moines, Iowa
  - University Health System: LSU Health Sciences, Shreveport, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Vascular Center, Flint, Michigan
  - Michigan Heart - St. Joseph Mercy Health System, Ypsilanti, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Rutgers University Hospital, Newark, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Mount Sinai Medical Center, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Greenville Memorial Hospital, Greenville, South Carolina
  - University of Virginia, Charlottesville, Virginia
  - Inova Heart and Vascular Institute, Falls Church, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Gunderson Health System, La Crosse, Wisconsin
  - University of Wisconsin - Madison, Madison, Wisconsin
- Canada (4):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences, Toronto, Ontario
  - Chu de Quebec, St-Francois d'Assise Hospital, Québec, Quebec
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
The proposed research will include data from approximately 500 subjects enrolled in the BEST-CLI clinical trial. The final dataset will include self-reported demographic, ultrasonographic, and laboratory data from the subjects. The investigators will be collecting identifying information, but the final dataset will be stripped of identifiers prior to release for sharing. Thus, the investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Sullivan AE, Huang S, Kundu S, Thomas VE, Clair DG, Aday AW, Menard MT, Farber A, Rosenfield K, Newman JD, Berger JS, Wells QS, Freiberg MS, Linton MF, Beckman JA. Association of Lipoprotein(a) With Major Adverse Limb Events and All-Cause Mortality Following Revascularization for Chronic Limb-Threatening Ischemia: A Substudy of the BEST-CLI Trial. J Am Heart Assoc. 2025 Jun 3;14(11):e041177. doi: 10.1161/JAHA.125.041177. Epub 2025 May 22. PMID 40401600